CLINICAL TRIAL: NCT06010654
Title: A Single Blind, Parallel Arm, Single Institution Pivotal RCT to Test Safety and Efficacy of Digital Therapeutics 'ANZEILAX' for Managing Generalized Anxiety Disorder
Brief Title: Pivotal RCT to Test Safety and Efficacy of Digital Therapeutics 'ANZEILAX' for Managing Generalized Anxiety Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: HAII corp.ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 3-2023-0018
Record Dates: First submitted 2023-08-20; First posted 2023-08-24 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Generalized Anxiety Disorder
MeSH Terms: conditions — Generalized Anxiety Disorder

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): The general treatment of the standard treatment method and the test device that provides self-talk training based on acceptance and commitment therapy (ACT) are used concurrently for 10 weeks.
  Interventions: Device: Software as a Medical device
- Control Group (No Intervention): Treatment as usual (TAU) is a standard treatment for 10 weeks, which is the clinical trial period.

INTERVENTIONS:
Device: Software as a Medical device — The test device is a software medical device designed for the purpose of treating generalized anxiety disorder that provides self-talk training based on acceptance and commitment therapy (ACT). Use 2 sets per day for 10 weeks with generalized treatment of standard treatment method.
  Other Names: ANZEILAX
  Arms: Experimental Group

SUMMARY:
The investigators propose to develop and adapt 'ANZEILAX' smartphone app specifically for individuals with Generalized anxiety disorder. The study will measure the therapeutic effects and safety of 'ANZEILAX' on symptoms of anxiety using pre- and post-treatment scores for generalized anxiety disorder and other physical, emotional, and cognitive symptoms of anxiety

DETAILED DESCRIPTION:
Purpose: This study is designed to evaluate the safety and efficacy of ANZEILAX, a digital therapeutic intervention delivered via a smartphone application. The application incorporates Acceptance and Commitment Therapy (ACT), a type of cognitive behavioral therapy, and self-communicational techniques to treat Generalized Anxiety Disorder(GAD). The study amis to assess the effectiveness to thie digital therapeutic in reducing anxiety symptoms and improving overall mental health outcomes in individuals with GAD.

Study Population: The study will enroll adults aged 19 years older who have completed at least a high school education.

Study Duration: The intervention period will last for 10 weeks, followed by a follow-up visit at Week 15 to assess long-term outcomes and effects after the completion of the intervention.

Intervention: Participants will use the smartphone application for a period of 10 weeks. The application is recommended to be used twice daily, with a minimum required use of once per day. It can be used during flexible time periods, such as before sleep, after waking up, or at any other when the participant feels it is necessary. The application delivers Acceptance and Commitment Therapy(ACT). It also encourages self-referencing activities, which help participants focus on and reflects upon experiences associated with positive emotions. Additionally, the application promotes self-distancing techniques, helping participants to avoid excessive immersion in negative emotional experiences.

ELIGIBILITY:
Inclusion Criteria:

People can participate in this clinical trial only if following criteria are met.

1. Adults aged 19 years or older with a high school diploma or higher
2. Disease groups according to the criteria below:

   * A person diagnosed with Generalized Anxiety Disorder (DSM-5 (ICD-10) code: 300.02 (F41.1))
   * Those who are classified as moderate or severe with 10 points or more through GAD-7
   * Those taking prescription drugs related to generalized anxiety disorder
3. A group of disorders with generalized anxiety disorder, or a group of disorders with worry that is a major symptom of generalized anxiety disorder in any of the following criteria:

   * Those suffering from other anxiety disorders such as panic disorder and social anxiety disorder
   * Those suffering from major depressive disorder accompanied by worry, the main symptom of generalized anxiety disorder
4. A person who fully understands the purpose, contents, and process of the clinical trial, agrees to participate, and signs the consent form in handwriting

Exclusion Criteria:

If any of the following criteria is applicable, the person cannot participate in this clinical trial.

1. Those who cannot read the consent form
2. Those who are inexperienced in using smartphones
3. In case of psychiatric symptoms or history (including schizophrenia, psychosis, bipolar disorder, epilepsy)
4. In case of brain damage, cognitive impairment, or neurological disease
5. In case of intellectual disability
6. Having a substance and alcohol use disorder
7. Suicidal intent, suicidal ideation, or self-injurious behavior in the past 6 months
8. Receiving cognitive behavioral therapy for anxiety, depression or mood disorders, or participating in such therapy in the past 3 months
9. Those who are registered in other clinical studies
10. Other investigators judged that the conduct of this clinical trial was inappropriate

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2023-08-14 (Actual); Primary Completion 2024-07-24 (Actual); Study Completion 2024-07-24 (Actual)

PRIMARY OUTCOMES:
Generalized Anxiety Disorder-7 | Measured at Baseline, Week 5, Week 10, and Week 15.
  The primary outcome will be measured using the Generalized Anxiety Disorder 7-item (GAD-7) scale, wich assesses the severity of generalized anxiety symptoms. The total score ranges from 0 to 21, with higher scores indicating more severe anxiety. Anxiety severity is categorized into four levels: 0-4(minimal anxiety), 5-9 (mile anxiety), 10-14 (moderate anxiety), and 15-21 (severe anxiety.)

SECONDARY OUTCOMES:
Beck Anxiety Inventory | Measured at Baseline, Week 5, Week 10, and Week 15.
  The Beck Anxiety Inventory (BAI) is a 21-tem, self-report tool designed to measure the severity of anxiety symptoms. It includes items that assess cognitive, emotional, and physical aspects of anxiety. The BAI is specifically designed to differentiate betwwen symptoms of ansiety and depression, with a focus on physical symptoms typically assocaiated with anxiety.
Penn State Worry Questionnaire | Measured at Baseline, Week 5, Week 10, and Week 15.
  The Penn State Worry Questionnaire (PSWQ) is a self-report tool developed to assess the presence and severity of pathologicla worry. It is designed to identify excessive, uncontrollabel worry, a key feafure of generalized anxiety disorder.
Hospital Anxiety and Depression Scale | Measured at Baseline, Week 5, Week 10, and Week 15.
  The Hospital Anxiety and Depression Scale(HADS) is a self-report tool used to assess anxiety symptoms, focusing on both physical and emotional aspects of anxiety. It is specifically designed for use in hospital settings to evaluate both anxiety and depression in patients.
Treatment adherence | Measured at Week 5 and Week 10
  During the clinical trial, Treatment As Usual (TAU) will vary depending on the severity of the participants' conditions, making it difficult to uniformly control across all subjects. Therefore, treatment adherence will be specifically assessed in the treatment group, where participants receive both TAU and ANZEILAX intervention. To evaluate adherence to the DTx, user log data from the DTx application will be collected and analyzed.
Satisfaction evaluation | Measured at Week 5 and Week 10
  Satisfaction with both Treatment As Usual (TAU) for anxiety and the digital therapeutic (DTx), ANZEILAX, will be assessed using two questions. The first question will ask participants to rate their satisfaction on a scale of 0 to 10, with 0 being "not satisfied" and 10 being "extremely satisfied." The second question will be an open-ended prompt asking participants to "write about their experiences during the treatment," allowing for qualitative feedback on their personal feelings and perceptions.

CONTACTS AND LOCATIONS:
Overall Officials: Jaejin Kim, Ph.D, Principal Investigator — Location Yonsei University Health System, Gangnam Severance Hospital
Locations (1):
- Yonsei University Health System, Gangnam Severance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Park C, Song H, Kim H, Kim E, Jo HJ, Kim JJ, Lee JH, Kim J. Efficacy of a Smartphone-Based Digital Therapeutic (Anzeilax) in Generalized Anxiety Disorder: Randomized Controlled Trial. J Med Internet Res. 2025 Oct 14;27:e69981. doi: 10.2196/69981. PMID 41086425